CLINICAL TRIAL: NCT05919212
Title: Trastuzumab Deruxtecan (T-DXd): Tailoring Treatment and Companion Diagnostics (CDx) by Liquid Biopsy. DIAMOND STUDY
Brief Title: Trastuzumab Deruxtecan (T-DXd): Tailoring Treatment and Companion Diagnostics (CDx) by Liquid Biopsy
Acronym: DIAMOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5382
Record Dates: First submitted 2023-05-18; First posted 2023-06-26 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with HER2 positive Breast cancer Stage IV (Experimental): All eligible patients to T-Dxd as second line treatment will receive T-Dxd intravenous at dose of 5,4 mg/kg every three weeks until progression disease or unacceptable toxicities.
  Subjects eligible to T-Dxd and who agree to participate in the study will undergo serial blood samples for liquid biopsy (LB) until progression disease.
  Interventions: Diagnostic Test: HER2-D is the use of a non-invasive liquid biopsy method to non-invasively and objectively assess HER2 status at recruitment

INTERVENTIONS:
Diagnostic Test: HER2-D is the use of a non-invasive liquid biopsy method to non-invasively and objectively assess HER2 status at recruitment — We study the circulating changes associated with resistance to T-DXd, including changes in HER2 status,studied through a new approach called HER2-2D that simultaneously assesses HER2 amplification and overexpression in blood

SUMMARY:
This is a prospective single-center pilot study phase II non randomized designed to explore the role of liquid biopsy in metastatic HER2-positive breast cancer patients treated with Trastuzumab deruxtecan (T-Dxd) as second line treatment according to international guidelines.

All eligible patients to T-Dxd as second line treatment will receive T-Dxd intravenous at dose of 5,4 mg/kg every three weeks until progression disease or unacceptable toxicities.

Subjects eligible to T-Dxd, who agree to participate in the study, will undergo serial blood samples for liquid biopsy (LB) until progression disease.

The timing of blood drawing will be scheduled as follows:

At each T-DXd administration for the first four cycles of T-Dxd (every three weeks). The next blood drawings will be done every three cycles of T-Dxd (every 9 weeks) until the thirteenth cycle. The next blood drawings will be done every six cycles of T-Dxd (every 18 weeks) until progression disease (documented by medical imaging) For all enrolled patients with available tumour tissue from primary diagnosis or last biopsy from recurrence, tissue samples will be requested for exploratory analysis.

DETAILED DESCRIPTION:
Human epidermal growth factor receptor 2-positive breast cancer represents 15%-20% of breast malignancies. In addition to this subtype characterized by HER2 overexpression or amplification, at least another 35% of breast cancer expresses HER2 at lower but detectable levels. These HER2-low tumors were defined as HER2 1+ and 2+ scores by immunohistochemistry (IHC) in the absence of gene amplification by in situ hybridization (ISH). There is evidence that HER2 overexpression/amplification may decrease during treatment HER2 blockade (4), determining that tumors of the 15% of HER2-positive group merge into the 35% of HER2-low group. Unfortunately, it is presently unclear how many HER2 overexpressing/amplified tumors are bound to join the HER2-low group, at which time during progression, and whether this may coincide to some extent with HER2 blockade inefficacy.

Traditionally, HER2 status is assigned: (a) at one point only (diagnosis), once and forever; (b) in tumor tissue only; (c) on a binary (yes/no) scale; and (d) with the limited aim of assigning conventional anti-HER2 therapy only. However, it is becoming increasingly clear that HER2 functional expression is not binary, but distributed along a continuum and intrinsically bimodal, e.g. (over)expression and copy number variations must be co-factored. It also appears that novel agents, such as Trastuzumab-deruxtecan (t-Dxd), may not be 'adapted' to the existing diagnostic scenario, but they may need a dedicated companion diagnostic (CDx). Moreover, IHC or ISH tissue diagnostic scheme is no longer applicable to the variety of available clinical HER2 blockade regimens and is in need of replacement. In this regard, liquid biopsy, with a comprehensive pan HER2 'unity solution', may be useful to capture HER2 on the wane as well as resistance traits, enable reallocation of patients to different subtypes, and assign treatment in a potentially practice-changing setting.

Preliminary data regarding the progressive HER2 loss during HER2 blockade and the potential of liquid biopsy in the metastatic HER-positive setting derive from the LiqBreasTrack trial (5). This is a small, single-center study exploring the role of liquid biopsy (at different time point from time zero until disease progression) in 22 HER2-positive breast cancer patients, treated with Trastuzumab emtansine (T-DM1) as per standard of care in 2nd or more line of therapy. Tumor DNA and circulating tumor DNA were tested by two commercial ThermoFisher targeted next generation sequencing (NGS) panels spanning about 50 (essentially overlapping) genes: the Ion AmpliSeqTM Cancer Hotspot and the OncomineTM Pan-Cancer panels. This study was designed to determine the potential impact of liquid biopsy in: 1) circulant tumor DNA (ctDNA) anticipation of clinical progression; 2. identification of recurrent mutational patterns on progression (e.g. alterations associated with, and possibly causative of, pharmacological resistance to T-DM1 and HER2 blockade altogether). The LiqBreasTrack trial showed that only five patients were still belonging to the 'HER2 subtype' (as assessed in blood) before T-DM1 administration. HER2 counterselection went on in all five of them, and a reversal to a HER2 neutral blood status was completed in the three who went all the way through >10 T-DM1 infusions until progression, whereas it was detectable, but incomplete, in the remaining two patients who had to discontinue T-DM1 due to rapid progression. Moreover, the development of a series of specific molecular alterations, either de novo appeared or progressively accumulated in blood, was associated (only when present in blood) with short time to progression. This suggests an oncogenic replacement of HER2 addiction by 'bypass' cancer drivers under strong and rapid adaptive selection pressure. This pilot study, although small, suggests several hypothesis: 1) T-DM1 (but this may apply to Trastuzumab-deruxtecan as well) rapidly pushes most or all tumors toward a presumably irreversible HER2 neutral state that had not been achieved by previous therapies; 2) in at least some cases, HER2-low tumors emerging from extensive HER2 blockade acquire features (e.g. hormone addiction) reminiscent of the naïve population of HER2-low tumors; 3) replacement of dominant HER2 addition comes at the cost (for the tumor) of developing alternative vulnerabilities, most of which had not been previously detected in tumor tissues, e.g. blood only alterations are the optimal biomarkers for cancer progression.

In summary, the HER2 loss may be a frequent event. It also remains to be determined how this HER2 loss intertwines with escape from HER2 blockade and the acquisition of the (so far scanty) list of adaptive resistance traits, both 'direct' (HER2 mutations) and 'bypass' (PTEN loss-of-function, PIK3CA mutations, integrin activation, YAP1 and IGF1 activation). In summary, regardless of whether constitutive or adaptively induced, an 'HER2-low status' spans a heterogeneous group of tumors comprising naïve and heavily pre-treated patients as well. Thus, there is an area of unmet medical need that may account for as many as 50% of all breast cancers and may include tumors on which neither conventional HER2 blockade nor hormone suppression strategies can determine a really clinical impact.

Liquid biopsy may reflect the dynamic changes in breast cancer biology, discriminate shades and grades of HER2 addiction and may be useful to identify the ideal CDx for Trastuzumab deruxtecan, the future second line standard of care for HER2-positive metastatic breast cancer (2). Indeed, liquid biopsy represents a non-invasive, non-dichotomic, quantitative, longitudinal test suitable for Trastuzumab-deruxtecan response monitoring and capturing potential mechanisms of resistance.

Based on these data, the DIAMOND study is a pilot, prospective study designed to primarily assess the ability of blood-based liquid biopsy using NGS to monitor disease progression to Trastuzumab-deruxtecan (as second line treatment) in patients with histologically confirmed diagnosis of HER2-positive metastatic disease previously treated with one treatment line for metastatic disease including pertuzumab with Trastuzumab or Trastuzumab alone (associated to taxane). The primary objective of the trial is to dynamically assess circulating alterations associated with resistance to Trastuzumab-deruxtecan, including changes of the HER2 status by a novel approach named HER2-2D that simultaneously assesses HER2 amplification and (over)expression in blood. The primary endpoint is the concordance between the clinical evaluation (progressive disease versus not progressive disease) based on RECIST criteria and the evaluation of liquid biopsy, (appearance of a new mutation and/or increasing of an existing one). Secondary objectives include: 1) molecular stratification of patients (dynamic approach by liquid biopsy); 2) lead time (anticipation of progression) assessment by liquid biopsy; 2) HER2-2D: use of a non-invasive liquid biopsy method to non-invasively and objectively assess HER2 status and to select patients displaying a HER2-low status.

Trastuzumab Deruxtecan will be administered at the dose of 5.4 mg per kilogram by intravenous infusion every 3 weeks (standard recommended dose). Treatment will be maintained until disease progression, severe toxicity or patient refusal. Liquid biopsy will be performed at baseline and repeated at different time points and/or at progression disease.

ELIGIBILITY:
Inclusion Criteria:

* Must be competent and able to comprehend, sign, and date informed consent prior to any study specific procedures;
* Male or female subjects age ≥ 18 years;
* Subjects with histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of either locally advanced disease not amenable to resection or radiation therapy with curative intent or metastatic disease not amenable to curative therapy;
* Subjects must have confirmed, per local testing on most recent tumor tissue sample available, an HER2-positive expression, as determined according to American Society of Clinical Oncology - College of American Pathologists guidelines (as defined in the 2013 American Society of Clinical Oncology (ASCO) recommendations for HER2 testing [7]) with any ER and/or PgR tumor status;
* Subjects must have received no more than one line of treatment including trastuzumab plus or not pertuzumab associated to taxane in the advanced/metastatic setting or progressed within 6 months after neoadjuvant or adjuvant treatment involving a regimen including trastuzumab and taxane;
* Documented radiologic progression (during or after most recent treatment or within 6 months after completing adjuvant therapy);
* Presence of at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (see Appendix A)
* Non measurable (evaluable) bone-only disease are eligible. Evaluable bone-only disease must include at least one lytic bone lesion or a mixed lytic-blastic bone lesion; blastic only metastases are not allowed. Subjects who have had prior radiation to bone must have at least one evaluable lesion in a non-irradiated area. Patients with lesions identified only on radionucleotide bone scan are not eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* Life expectancy > 12 weeks;
* Subjects with clinically inactive brain metastases may be included in the study.
* Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of brain radiotherapy and study enrolment.
* LVEF ≥ 50% within 28 days before enrolment.
* Adequate organ and bone marrow function within 14 days before enrollment
* Adequate treatment washout period before enrolment
* Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of IMP. Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause.
* Agree for periodically blood sample collection for liquid biopsy

Exclusion Criteria:

* Prior treatment with an anti-HER2 Antibody Drug Conjugated (ADC)
* Uncontrolled or significant cardiovascular disease, including any of the following:

  a. History of myocardial infarction (MI) within 6 months before enrolment; b. History of symptomatic congestive heart failure (New York Heart Association Class II to IV); c. Corrected QT interval (QTc) prolongation to > 470 ms (females) or >450 ms (male) based on average of Screening triplicate 12-lead ECG; d. Left ventricular ejection fraction (LVEF) < 50% within 28 d prior to enrollment
* History of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
* Lung criteria: a. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrolment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.); b. Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study; c. Prior pneumonectomy (complete)
* Spinal cord compression or clinically active central nervous system (CNS) metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
* Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects should be tested for HIV prior to enrolment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
* Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of T-Dxd. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study treatment.
* Multiple primary malignancies within 3 years, except adequately resected non melanoma skin cancer, curatively treated in situ disease, other solid tumors curatively treated, or contralateral breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Alterations associated with resistent to Trastuzumab Deruxtecan | 4 years
  To dynamically assess circulating alterations associated with resistance to Trastuzumab Deruxtecan (T-DXd) including changes of the HER2 status by a novel approach named HER2-2D that simultaneously assesses HER2 amplification and (over)expression in blood.

SECONDARY OUTCOMES:
Molecular stratification of patients (dynamic approach by Liquid Biopsy, LB); | 4 years
  Listing of circulating alterations during treatment and at progression: particularly those actionable at OncoKB level 3A/B or lower, particularly when ctDNA-only
Lead Time assessment by Liquid Biopsy. | 4 years
  LB Lead Time Progression Free Survival (PFS-LB) compared to medical imaging, Lead Time is defined as the time to progression by RECIST.1 criteria (PFS-R) - (minus, subtraction) the time to progression by circulating tumor DNA, e.g. PFSctDNA. Days of Lead Time= days PFS-R - days PFS-ctDNA
Association between HER2-2D and outcome in terms of progression. | 4 years
  PFS assessed between two groups of patients in relation with HER2-2D: HER2 status lower vs higher detected by LB.

OTHER OUTCOMES:
To evaluate the safety and tolerability of T-Dxd | 4 years
  Toxicity will be graded according to NCI-CTCAE vers. 5.0
To evaluate the concordance or not between mutations discovered at baseline liquid biopsy and tissue extraction mutations from primary or last available tumor tissue | 4 years
  To assess whether the presence of tissue genomic alterations found in liquid biopsy are comparable to those identified in neoplastic tissue (from primary tumor tissue or the last available tumor tissue) and whether they are associated and with drug resistance and susceptibility to T-DXd

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Fondazione Policlinico A. Gemelli - IRCCS
Locations (1):
- Fondazione Policlinico A. Gemelli - IRCCS, Rome, Italy